CLINICAL TRIAL: NCT01628978
Title: Verification of Appropriate Insertion Depth of Endotracheal Tube Placement in Infants and Young Children by Ultrasonography
Brief Title: Verification of Appropriate Insertion Depth of Endotracheal Tube Placement
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Sangmin M. Lee, Professor, Samsung Medical Center
Other Study IDs: 2012-05-028-001
Record Dates: First submitted 2012-06-24; First posted 2012-06-27 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Endotracheal Intubation; Infants or Young Children
Keywords: depth of endotracheal tube placement; endotracheal intubation; endobronchial intubation
MeSH Terms: interventions — Auditory Perception

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Auscultation group: The depth of endotracheal tube placement is determined by auscultation.
  Interventions: Other: determination by auscultation
- Ultrasonography group: The depth of placement of endotracheal tube placement is determined by ultrasonographic finding of pleural sliding sign.
  Interventions: Other: determination by ultrasound

INTERVENTIONS:
Other: determination by auscultation — determination of depth of endotracheal tube placement by auscultation
  Other Names: auscultation
  Groups: Auscultation group
Other: determination by ultrasound — determination of depth of endotracheal tube placement by ultrasound
  Other Names: H-Universal Stand (sonosite, Bothell, WA, USA)
  Groups: Ultrasonography group

SUMMARY:
The investigators are trying to evaluate the efficacy of ultrasonographic determination of depth of endotracheal tube placement in infants and young children by using the pleural sliding sign.

DETAILED DESCRIPTION:
It is difficult to determine the adequate depth of endotracheal tube placement in infants and young children. It is usually determined by an equation according to the patient's age (12 + age/2, cm) or auscultation method. The auscultation method is to intentionally place the tip of the endotracheal tube into the right main stem bronchus and then withdraw it until breath sounds are equal. The tube is fixed 1 or 2 cm proximal to the point where breath sounds become equal. However, in small children or infant, as the breadth sound in unilateral lung transmits the contralateral lung field and is often difficult to listen in a noisy operation room, it is often difficult to determine the depth by auscultation method. Pleural sliding sign, or sliding lung sign is a ultrasonographic finding that the visceral pleura moves against the parietal pleura. It is used to identify whether the lung is ventilated by ultrasound. The investigators are trying to use this pleural sliding sign to determine the depth of endotracheal tube, and compare this method with auscultation method.

ELIGIBILITY:
Inclusion Criteria:

* Infants or young children (less than body weight of 20 kg) undergoing elective surgery (general surgery, urology, plastic surgery, cardiac surgery) under general anesthesia with endotracheal intubation

Exclusion Criteria:

* Patients with pneumothorax, pleural effusion, atelectasis, pneumonia
* hemodynamic unstable patients (inotropics use)
* History of difficult intubation
* Combined upper airway anomaly

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants or young children (less than body weight of 20 kg) undergoing elective surgery (general surgery, urology, plastic surgery, otolaryngologic surgery, cardiac surgery) under general anesthesia with endotracheal intubation
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
the incidence of inadequate depth of endotracheal tube placement by flexible brochoscopy after intubation | 3 minutes after intubation
  the incidence of inadequate depth of endotracheal tube placement by flexible bronchoscopy 3 minute after intubation

SECONDARY OUTCOMES:
incidence of repositioning of endotracheal tube placement | 10 min after anesthetic induction
  incidence of repositioning of endotracheal tube placement (when it is found that the depth of endotracheal tube placement was inadequate determined by saturation fall or airway pressure monitoring)
time to verification of appropriate insertion depth of endotracheal tube placement | 30 minutes after the end of surgery
  time to verification of appropriate insertion depth of endotracheal tube placement by a independent observer
blood pressure | 5, 10, 20 min after anesthetic induction
  systolic, diastolic, mean blood pressure before attempt of endotracheal intubation (5 min), during determining the depth of endotracheal tube placement (10 min), after determining the depth of endotracheal tube placement (20 min)
heart rate | 5, 10, 20 min after anesthetic induction
  heart rate before attempt of endotracheal intubation (5 min), during determining the depth of endotracheal tube placement (10 min), after determining the depth of endotracheal tube placement (20 min)
pulse oximetry | 5, 10, 20 min after anesthetic induction
  pulse oximetry before attempt of endotracheal intubation (5 min), during determining the depth of endotracheal tube placement (10 min), after determining the depth of endotracheal tube placement (20 min)

CONTACTS AND LOCATIONS:
Overall Officials: Sangmin M. Lee, MD, PhD, Principal Investigator — Samsung Medical Center; Won Ho Kim, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea